CLINICAL TRIAL: NCT05473169
Title: Evaluation of Swallowing in Patients With Vocal Folds Immobility
Brief Title: Swallowing Evaluation in VF Immobility
Status: Unknown | Type: Observational
Last Known Status: Not yet recruiting
Sponsor: Assiut University (Other)
Responsible Party: Principal Investigator, Mohamed Zakaria Ahmed Elbakry, Principal investigator, Assiut University
Other Study IDs: Swallowing in VF immobility
Record Dates: First submitted 2021-12-21; First posted 2022-07-25 (Actual); Last update posted 2022-07-25 (Actual); Status verified 2022-07

CONDITIONS: Swallowing Disorder
MeSH Terms: conditions — Deglutition Disorders

STUDY DESIGN:
Observational Model: Case-Control | Time Perspective: Cross-Sectional
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (2):
- Patients: Patients with Vocal fold immobility
  Interventions: Device: Videofluoroscopy
- Control: Normal volunteer don't have dysphagia , neurological diseases , heart burn and acid regurgitation
  Interventions: Device: Videofluoroscopy

INTERVENTIONS:
Device: Videofluoroscopy — Swallowing assessment
  Other Names: Nasofibroscopy

SUMMARY:
Vocal fold immobility (VFI) often results in significant problems with dysphonia, dysphagia, and decreased cough strength. As one element of the dysphagia potentially associated with vocal fold immobility,

aspiration may create significant morbidity for these patients. An estimated 38% to 53% of patients with

untreated VFI have swallowing difficulties with aspiration.

Vocal fold immobility has important implication on the laryngeal airway protection during respiration,

phonation and swallowing. It is the most common neurological laryngeal disorder.

The immobility may be caused by neck and thoracic surgery. which can impair the innervation of the pharynx,

upper esophageal sphincter (U.E.S) and proximal esophagus but may also be due to malignancy,trauma,

Intracranial causes,or may be idiopathic

DETAILED DESCRIPTION:
Besides the voice alteration, the lesion that causes of vocal fold immobility should also affect the pharyngeal phase of swallowing.

It was suggested that dysphagia in patient with vocal fold immobility has multifactor causes ; including limited airway protection and decrease laryngopharyngeal sensation based on the finding of the flexible endoscopy.

Another study revealed that pharyngeal phase abnormalities such as delayed initiation of swallowing, reduced laryngeal elevation, and reduced upper esophageal sphincter (UES) opening were found in video fluoroscopic swallowing studies (VFSS).

Several studies on the swallowing difficulties of patient with vocal fold immobility has been performed and reported that nearly 56% of these patients immobility have swallowing dysfunction.

ELIGIBILITY:
Inclusion Criteria:

1. Age:above 18.
2. Gender:both sexes will be included in the study.

Exclusion Criteria:

1. patients with structural abnormalities of oral cavity, pharynx or larynx.
2. previous vocal fold injection or voice therapy.
3. other causes of dysphagia: esophageal cancer or spasm , gastric cancer, cancer larynx,or radio therapy .
4. . Patients with history of heart burn , acid regurgitation ,
5. other neurological disease ,stroke, hypothyroidism or dyspnea.

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Study Population: Patients with Vocal fold immobility
Sampling Method: Probability Sample
Enrollment: 40 (Estimated)
Dates: Start 2022-07 (Estimated); Primary Completion 2023-07 (Estimated); Study Completion 2023-08 (Estimated)

PRIMARY OUTCOMES:
To calculate the incidence of swallowing dysfunction in people with vocal fold immobility | Baseline
  Incidence of swallowing dysfunction in patients with vocal fold immobility will be determined by the Statistical Package for the Social Sciences (SPPS) after the diagnosis of swallowing dysfunction by fiberoptic endoscopic evaluation of swallowing (FEES) and videofluoroscopic swallow study (VFSS)

SECONDARY OUTCOMES:
Measure the frequency of each swallowing phase which will be affected in vocal fold immobility patients | Baseline
  To detect which swallowing phase is causing the dysfunction by using Statistical Package for the Social Sciences (SPSS) program

CONTACTS AND LOCATIONS:
Overall Officials: Assiut, Principal Investigator — Non-afiliated

IPD SHARING:
Plan to Share IPD: Undecided
Undecided

REFERENCES:
- [Background] Heitmiller RF, Tseng E, Jones B. Prevalence of aspiration and laryngeal penetration in patients with unilateral vocal fold motion impairment. Dysphagia. 2000 Fall;15(4):184-7. doi: 10.1007/s004550000026. PMID 11014880
- [Background] Ollivere B, Duce K, Rowlands G, Harrison P, O'Reilly BJ. Swallowing dysfunction in patients with unilateral vocal fold paralysis: aetiology and outcomes. J Laryngol Otol. 2006 Jan;120(1):38-41. doi: 10.1017/S0022215105003567. Epub 2005 Nov 25. PMID 16359143